CLINICAL TRIAL: NCT04361240
Title: Cardiotoxicity in Breast Cancer Patients Treated With Proton or Photon Radiotherapy: A RadComp Companion Study
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UPCC 17119
Record Dates: First submitted 2020-04-06; First posted 2020-04-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Cardiotoxicity
Keywords: Cardio-Oncology; Radiation Therapy Cardiotoxicity
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, and Buffy coat are collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary Cohort: No Intervention: Subjects will be followed before, during and for up to 1 year after radiation with echocardiogram, blood draw, and symptoms and activity survey.
  Interventions: Radiation: Proton vs Photon Radiation

INTERVENTIONS:
Radiation: Proton vs Photon Radiation — Assignment to proton vs photon by randomization on RadComp parent study.

SUMMARY:
This is a companion study to the "Pragmatic Randomized Trial of Proton vs Photon Therapy for Patients with non-Metastatic Breast Cancer Receiving Comprehensive Nodal Radiation: A Radiotherapy Comparative Effectiveness (RadComp) Consortium Trial" (NCT02603341). The investigators will collect cardiovascular (CV) biomarkers and echocardiograms prior to, during, and for up to 1 year following radiation for a subset of patients enrolled on RadComp and to evaluate the impact of proton vs photon radiation therapy (RT) on CV function and structure.

DETAILED DESCRIPTION:
The study population of the companion study will consist of newly enrolled RadComp trial participants. Patients on this ancillary will be consented prior to RadComp randomization to decrease the bias secondary to RT type and enhance internal validity. The study will define the early changes in biomarkers, imaging measures, and RT dose volume metrics and long-term (5-10 year) CV clinical outcomes using the RadComp parent study's infrastructure for clinical data collection and long-term follow-up. Blood samples, echocardiograms, and questionnaires are obtained at baseline (between end of chemotherapy and start of RT), immediately after the end of RT, and at 6 months and 12 months after the end of RT. An additional blood sample will be collected at 4 weeks after the start of RT. Clinical, demographic, and patient reported outcomes data are collected as part of the RadComp parent study. In addition to data collected by RadComp, we will collect a limited set of clinical data and two additional quality of life instruments for the companion study.

ELIGIBILITY:
Inclusion Criteria:

* Consented to RadComp
* Willing and able to provide written consent

Exclusion Criteria:

* Knowledge of randomization on RadComp prior to enrollment on companion study
* Non-diagnostic echocardiography windows as assessed on local read.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for and enrolling on the RadComp trial at participating RadComp sites will be approached for the companion cohort.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 14 months
  Change in echocardiography derived LVEF from baseline
Right Ventricular (RV) Fractional Area Change (FAC) | 14 months
  Change in echocardiography derived RV FAC from baseline
Circulating N-terminal pro B-type natriuretic peptide (NTproBNP) | 14 months
  Change in NTproBNP levels from baseline
Circulating Placental Growth Factor (PIGF) | 14 months
  Change in PIGF levels from baseline
Circulating Growth Differentiation Factor-15 (GDF-15) | 14 months
  Change in GDF-15 levels from baseline

SECONDARY OUTCOMES:
LV systolic strain | 14 months
  Change in 2D echocardiography derived LV global longitudinal strain and circumferential strain from baseline
Echocardiography derived Ventricular Arterial Coupling Measurement | 14 months
  Change from baseline in ventricular arterial coupling as defined by end systolic elastance divided by effective arterial elastance
Diastolic function (E/e') | 14 months
  Change in E/e' from baseline as measured by echocardiogram
Circulating Troponin T(TnT) | 14 months
  Change in high-sensitivity TnT levels from baseline
Circulating high-sensitivity C-Reactive Protein (hsCRP) | 14 months
  Change in hsCRP levels from baseline

OTHER OUTCOMES:
3D LVEF | 14 months
  Change in 3d echocardiography derived LVEF from baseline
3D LV systolic strain | 14 months
  Change in 3D echocardiography derived longitudinal and circumferential strain from baseline
LV Twist and Torsion | 14 months
  Change in 3D echocardiography derived measures of LV twist and torsion from baseline
Patient Reported Outcomes (PRO) Common Terms and Criteria for Adverse Events (CTCAE) | 14 months
  Incidence and severity of PRO CTCAEs
Incidence of major cardiovascular events (MCE) | 10 years
  Collected, defined, and adjudicated by the RadComp study team

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Ky, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Alabama
  - Northwestern Medicine, Warrenville, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided
Participants may opt in to allowing data and/or banked samples to be used for future research and shared with other researchers. A detailed plan for sharing IPD will be finalized at a later date, and may depend in part on how many participants elect this option. Additional supporting information may be shared, including the study protocol and informed consent form.